CLINICAL TRIAL: NCT00472563
Title: Prevention of Contrast Induced Nephropathy With Sodium Bicarbonate
Acronym: PROMEC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 065-120606
Record Dates: First submitted 2007-05-10; First posted 2007-05-11 (Estimated); Last update posted 2008-05-06 (Estimated); Status verified 2008-04

CONDITIONS: Acute Kidney Failure
Keywords: bicarbonate; nephropathy; contrast
MeSH Terms: conditions — Acute Kidney Injury; Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Bicarbinate 150 mEq/L — 75 cc of sodium bicarbonate (8.4%) mixed in 425 cc of D5W

SUMMARY:
Deterioration of kidney renal function occurs in a minority of people due to contrast-required procedures. The purpose of this study is to compare two different interventions to reduce the risk of kidney injury after contrast medium exposition.

We will perform a randomized clinical trial following a modification of a previously published protocol (Merten et al.JAMA 2004;291(19):2328-34). Patients will be randomly assigned to one of two groups of treatment. Group A will receive 1 cc/kg/hour of 0.9% saline infusion starting 12 hours before and continuing 12 hours after the procedure. Group B will receive 3 cc/kg of sodium bicarbonate solution for one hour prior to procedure, then drip rate will be decreased to 1 cc/kg/hour until 6 hours post procedure.

DETAILED DESCRIPTION:
We will perform a randomized clinical trial following a modification of a previously published protocol (Merten et al.JAMA 2004;291(19):2328-34). Patients will be randomly assigned to one of two groups of treatment. Group A will receive 1 cc/kg/hour of 0.9% saline infusion starting 12 hours before and continuing 12 hours after the procedure. Group B will receive 3 cc/kg of sodium bicarbonate solution for one hour prior to procedure, then drip rate will be decreased to 1 cc/kg/hour until 6 hours post procedure.

Phase 2/3 study Study Type: Interventional Study Design: Prevention, Randomized, Open Label, Active Control, Parallel Assignment, Efficacy Study.

Subjects: Consecutive samples of all inpatients who meet the inclusion criteria

Primary outcomes: Development of contrast induced nephropathy, defined as an increase in serum creatinine of 25% or more within 48 h after administration of contrast.

Secondary outcomes: change in serum bicarbonate; change in serum potassium; change in serum creatinine.

Expected total enrollment: 212

Allocation Assignment: Patients who meet inclusion criteria and agree to participate in the study will be assigned by a random number table to saline or bicarbonate, using closed envelopes and stratifying according to history of diabetes and type of procedure (cardiac catheterism or others).

Condition: Contrast Induced Nephropathy

Intervention: 75 cc of sodium bicarbonate (8.4%) mixed in 425 cc of D5W

Gender: both Age: 18+ years of age Recruitment Status: participants are currently being recruited

Facility location:

Universidad de Antioquia, Internal Medicine Department; Hospital Universitario San Vicente de Paul. Medellin, Colombia.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* Inpatient at Hospital Universitario San Vicente de Paúl scheduled to undergo diagnostic CT scan using contrast or angiography and either

  * Serum creatinine 1.2 mg/dl or more, or
  * Type 2 Diabetes Mellitus

Exclusion Criteria:

* Current clinical diagnosis of exacerbated congestive heart failure
* Exposure to contrast 30 days prior to study
* Allergy to contrast dye
* Chronic renal disease with dialysis therapy
* Acute renal failure with dialytic urgency
* Urgency procedure needed
* Systolic blood pressure < 90 or vasopressor support
* No authorization by patient or physician in charge
* Serum potassium < 3 mEq/L
* Ejection fraction < 35% by previous echocardiography
* Acute pulmonary edema in previous 48 hours

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2007-05; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
development of contrast induced nephropathy, defined as an increase in serum creatinine of 25% or more within 48 h after administration of contrast | 48 h

SECONDARY OUTCOMES:
change in serum bicarbonate; change in serum potassium; change in serum creatinine | 48 h

CONTACTS AND LOCATIONS:
Overall Officials: Wilmar A Maya Salazar, MD, Principal Investigator — Universidad de Antioquia; Julián M Aristizábal, MD, Study Chair — Universidad de Antioquia; Oscar M Santos, MD, Study Chair — Universidad de Antioquia; John F Nieto, MD, Study Chair — Universidad de Antioquia; Liliana Jaramillo, MD, Study Chair — Universidad de Antioquia; Jorge I García, MD, Study Chair — Universidad de Antioquia; Fabian A Jaimes, MD, Study Director — Universidad de Antioquia; Alvaro García, MD, Study Chair — Universidad de Antioquia
Locations (1):
- Hospital Universitario San Vicente Paúl, Medellín, Antioquia, Colombia